CLINICAL TRIAL: NCT00545493
Title: Efficacy of Tacrolimus and i.v.-Immunoglobulins in Rasmussen Encephalitis With Start of Treatment in the Acute Disease Stage. Prospective, Randomised, Open Parallel Group Study
Brief Title: Efficacy of Tacrolimus and I.V.-Immunoglobulins in Rasmussen Encephalitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: Octapharma (Industry); Astellas Pharma GmbH (Industry)
Responsible Party: PD Dr. Christian G. Bien, MD, University of Bonn, Dept. of Epileptology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 135/02
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2009-04-10 (Estimated); Status verified 2009-04

CONDITIONS: Rasmussen Encephalitis
Keywords: Rasmussen encephalitis; Chronic encephalitis; Cerebral hemiatrophy; Hemiparesis; Epilepsy
MeSH Terms: conditions — Encephalitis; Paresis; Epilepsy | interventions — Tacrolimus; Octagam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Tacrolimus capsules ("Prograf"; dosing according to blood trough levels: 12-15 ng/ml during months 1-6, 5-10 ng/ml during months 7-12 and 5-8 ng/ml thereafter)
  Interventions: Drug: Tacrolimus
- Group 2 (Experimental): Intravenous immunoglobulins (IVIG) infusions ("Octagam"; dosing: initially on three consecutive days 0,4 g/kg KG, thereafter 0,4 g/kg KG every month, after 12 months of treatment every two months).
  Interventions: Drug: i.v. immunoglobulins

INTERVENTIONS:
Drug: Tacrolimus — tacrolimus capsules, dosing according to blood trough levels: 12-15 ng/ml during months 1-6, 5-10 ng/ml during months 7-12 and 5-8 ng/ml thereafter
  Other Names: Prograf
  Arms: Group 1
Drug: i.v. immunoglobulins — infusions, dosing: initially on three consecutive days 0,4 g/kg KG, thereafter 0,4 g/kg KG every month, after 12 months of treatment every two months).
  Other Names: Octagam
  Arms: Group 2

SUMMARY:
Rasmussen encephalitis (RE) is a rare but severe chronic inflammatory brain disease of unknown origin affecting one brain hemisphere. It is usually accompanied by intractable epilepsy. In addition, it often leads to severe disability due to functional deficits caused by atrophy of one brain hemisphere. Hemispherectomy is an effective means of surgical treatment of the epilepsy. It renders the patient, however, hemiplegic, hemianopic and (if the language dominant hemisphere is affected) aphasic. To slow down or even stop the progressive inflammatory damage to the affected brain hemisphere, immunotherapies may be beneficial. According to a literature survey, tacrolimus (twice daily intake of capsules) and intravenous immunoglobulins (monthly infusions) are the most promising compounds for this. In the investigators' study, these two types of treatment are randomly assigned to patients with disease onset within the last year and not too far advanced disability or hemispheric brain injury. The patients are followed to assess prospectively the functional and brain MRI course of the disease.

DETAILED DESCRIPTION:
1. Trial design/2. Trial interventions Patients are screened in epileptological, neuropediatric, and neurological centers all over Germany. The study design was approved on a meeting in Bonn on April 20, 2002 by several external participants and by the ethical committee of the University of Bonn. Patients with the suspected diagnosis of RE are transferred to the Department of Epileptology of the University of Bonn. If the diagnosis "RE in the acute stage" is confirmed and the patient or (in children) the parents give informed consent, the patients are randomized to one of the two active treatment arms.

The study was started on 1.10.2002. The first patient was included on 20.11.2002.

3. Inclusion/exclusion criteria See appropriate section

4. Duration Recruitment started on 1.10.2002 and will go on until the proposed number of study participants has been included. A patient remains in the study until he or she reaches one of the predefined exit parameters (see below, #4.5). Every patient will be followed under study conditions for at least 12 months (to obtain true long term results).

5. Outcome measures See appropriate section.

6. Methods against bias The patients will be randomized to one of the treatment arms. To avoid unbalanced group sizes and unequal numbers of adolescents and adults, there are two randomization lists, one for patients < 11 years, one for older patients (stratification). Blinding is not possible because the administration of the two drugs is different and would have necessitated the additional use of placebo capsules in the IVIG group and placebo infusions in the tacrolimus group. Because the production and administration of an adequate "IVIG-placebo" is highly impracticable, no blinded treatment application was planned. The physicians assessing the "Motricity Index" and the "Hemispheric ratio" are unaware of the kind of treatment used.

7. Power calculations It is assumed that 1-2 RE patients are diagnosed at a large epilepsy center per year. The cooperation of the study center with the other specialized centers in Germany is good. Therefore, it is expected that the majority of RE cases are transferred to or department. We estimated that 16 suitable patients can be included within the proposed inclusion period. The disease is too rare to perform power calculations (which are mainly used to limit recruitment figures). RE is an orphan disease, so even if the number of participants will not suffice to detect small to moderated differences between the two treatments, the results will provide invaluable information on the conservative treatment of the condition, e.g. in comparison to historical untreated controls.

8. Number of participants It is intended to include at least 16 patients during the above named period (otherwise, the recruitment period will be prolonged). We will perform an intention to treat analysis and an analysis of the patients treated per protocol.

9. Trial sites Potential study participants are referred to our department (Dept. of Epileptology, University of Bonn) from all over Germany. The study procedures, especially the clinical and neuroradiological follow-up studies including assessment of safety parameters are performed in Bonn (visits every two months within the first year, in the second year every four months, thereafter every six months). In the intervals between the visits in Bonn, the referring centers participate in monitoring of the patients and administration of IVIG. There is continuous contact between the study center Bonn and the external study co-workers.

10. Analyses Primary outcome parameter (time to exit): The two groups will be compared by the log rank test (Kaplan-Meyer-survival curves). Non-parametric tests will be applied for the secondary outcome parameters.

11. Ethical considerations Tacrolimus and IVIG can have side effects. The known tacrolimus side effects are more severe and more frequent than those of IVIG. It must be noted, however, that the known tacrolimus side effects were assessed in organ transplant patients who had severe medical diseases and were usually treated with more than one immunosuppressant. In patients with autoimmune disorders treated with tacrolimus-monotherapy, the side effects were considerably lower. RE itself is a disease with a deleterious natural course so that the possible risks of an immunotherapy are clearly outweighed. It must be assumed that most RE patients worldwide are treated with any kind of immunotherapy in the early disease stage due to the favorable case reports in the literature. Therefore, a placebo control group appears ethically unacceptable. This is why we chose to compare the two most promising substances. The ethics committee of the University of Bonn has approved the study design.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting at least two of the following three criteria:

  1. Clinical: Epilepsia partialis continua or progressive* hemiparesis
  2. MRI: Progressive* cerebral hemiatrophy
  3. Histopathology: T cell dominated encephalitis with activated microglial cells (typically, but not necessarily forming nodules) and reactive astrogliosis. Numerous macrophages, B cells or plasma cells or positive signs of viral infections (viral inclusion bodies or immunohistochemical demonstration of viral protein) exclude the diagnosis of RE.

     * "Progressive" means that at least two sequential clinical examinations or MRI studies documenting increasing deficits or tissue loss are required to meet the respective criteria.

Exclusion Criteria:

* Neuroradiological signs of a bihemispheric encephalitis.
* Wave-like course with history of repeated remissions.
* Infectious disease as a contraindication to an immunosuppressive therapy.
* Paraneoplastic encephalitis.
* Previous treatment with > 3 weeks of corticosteroids or tacrolimus or > 1,2 g/kg IVIG or > 5 PEX/PAI within the last three months.
* Onset of acute disease stage more than 12 months ago.
* Patient already in residual stage, i.e., stable neurological deficit since >6 months.
* Hemispheric Ratio < 80% (< 90% in patients > 11 years)
* Histopathological evidence of cerebral inclusion bodies indicating a viral infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2002-11; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Time to exit, criteria: Deterioration of motor function of the affected side by 15 % (>11 yrs of age: 8%) measured by the "Motricity Index" (scale 0-100) or deterioration of the "Hemispheric ratio" assessed by regular MRI scans by 15% (>11 yrs: 8%). | until final included subject has been followed for one yer

SECONDARY OUTCOMES:
seizure frequency, "Burden of disease" scale, neuropsychological performance, quality of life, T cell receptor studies (H Wiendl, Würzburg) | until final included subject has been followed for one yer

CONTACTS AND LOCATIONS:
Overall Officials: Christian G Bien, M.D., Principal Investigator — University Hospital Bonn, Bonn, Germany
Locations (1):
- University of Bonn, Dept. of Epileptology, Bonn, Germany

REFERENCES:
- [Background] Bien CG, Gleissner U, Sassen R, Widman G, Urbach H, Elger CE. An open study of tacrolimus therapy in Rasmussen encephalitis. Neurology. 2004 Jun 8;62(11):2106-9. doi: 10.1212/01.wnl.0000128044.94294.87. PMID 15184626
- [Background] Bien CG, Granata T, Antozzi C, Cross JH, Dulac O, Kurthen M, Lassmann H, Mantegazza R, Villemure JG, Spreafico R, Elger CE. Pathogenesis, diagnosis and treatment of Rasmussen encephalitis: a European consensus statement. Brain. 2005 Mar;128(Pt 3):454-71. doi: 10.1093/brain/awh415. Epub 2005 Feb 2. PMID 15689357
- [Background] Granata T, Fusco L, Gobbi G, Freri E, Ragona F, Broggi G, Mantegazza R, Giordano L, Villani F, Capovilla G, Vigevano F, Bernardina BD, Spreafico R, Antozzi C. Experience with immunomodulatory treatments in Rasmussen's encephalitis. Neurology. 2003 Dec 23;61(12):1807-10. doi: 10.1212/01.wnl.0000099074.04539.e0. PMID 14694056
- [Background] Hart YM, Cortez M, Andermann F, Hwang P, Fish DR, Dulac O, Silver K, Fejerman N, Cross H, Sherwin A, et al. Medical treatment of Rasmussen's syndrome (chronic encephalitis and epilepsy): effect of high-dose steroids or immunoglobulins in 19 patients. Neurology. 1994 Jun;44(6):1030-6. doi: 10.1212/wnl.44.6.1030. PMID 8208394
- See also: Homepage of institution performing the trial — http://www.meb.uni-bonn.de/epileptologie/cms/front_content.php?changelang=3